CLINICAL TRIAL: NCT05678439
Title: Effects of Sesamin on Sleep Quality and Antioxidative Status in Low Arousal Threshold Obstructive Sleep Apnea Syndrome Patients and Patients With Risk of Obstructive Sleep Apnea Syndrome
Brief Title: Effects of Sesamin on Sleep Quality and Antioxidative Status
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Taipei Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Prevention
Other Study IDs: N202205061
Record Dates: First submitted 2022-10-02; First posted 2023-01-10 (Actual); Last update posted 2024-05-23 (Actual); Status verified 2023-10

CONDITIONS: Sleeping Disorders
Keywords: Sleeping Disorders; sesamin; antioxidant
MeSH Terms: conditions — Parasomnias

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- sesame extract (Experimental): Dietary supplement: sesame extract (contains sesamin 37-56mg per capsule)
  This group will be given supplements for 8 weeks.
  Interventions: Dietary Supplement: sesame extract
- placebo (Placebo Comparator): Placebo treatment ( identical capsules containing Lactose, Silica, Magnesium Stearate, Gelatin)
  Interventions: Other: placebo

INTERVENTIONS:
Dietary Supplement: sesame extract — At the treatment period (0th to 8th week of the experiment), participants with sleeping disorder will receive 2 capsules of sesame extract (sesamin 37-56mg per capsule). The 8th to 9th week will be the washout period. The placebo group and sesame extract group will be cross-over at 10th week to 18th week of the experiment.
  Arms: sesame extract
Other: placebo — At the treatment period (0th to 8th week of the experiment), participants with sleeping disorder will receive 2 capsules of placebo. The 8th to 9th week will be the washout period. The placebo group and sesame extract group will be cross-over at 10th week to 18th week of the experiment.
  Arms: placebo

SUMMARY:
Sesame recognized as a common healthy food. Sesamin is extracted from sesame and has high antioxidant capacity which is commonly added in functional foods. Present studies had found sesamin supplementation could improve self-reported fatigue but more evidence should be clarify. The purpose of this study is to evaluate the effects of sesame extract on the quality of life and antioxidative status on sleeping disorder patients with not or with low arousal threshold obstructive sleep apnea and assess the potential product development.

DETAILED DESCRIPTION:
30-50 subjects aged from 20 to 80 years old without sleep apnea or with low arousal threshold obstructive sleep apnea will be enrolled in this randomized, double-blind, cross-over, and placebo-controlled 8-week period experiment.

At the treatment period (0th to 8th week of the experiment), subjects will receive 2 placebo or capsules of sesame complex (37-56mg sesamin per capsule). The 9th to 11th week will be the washout period. The control and sesamin group will be cross-over at 11th week to 12th week of the experiment. Sleep quality, life quality examination and anti-oxidative functions will be carried out in this study. The basic anthropometric examination will be carried out at the beginning, 4th, 8th, 11th, 15th, and 19th week of the study. Routine laboratory parameters including liver function, kidney function, blood sugar, lipid profile, and anti-oxidative status will be investigated at the beginning, 8th, 11th and 19th week of the study. The questionnaire evaluation including the Pittsburgh Sleep Quality Index, Epworth Sleepiness Scale, Beck Depression Inventory-II, Beck Anxiety Inventory, and Short form-12 items health survey will be investigated at the beginning, 8th, 11th, and 19th week of the study. We expect that sesame complex including 37-56mg sesamin may improve oxidative status which in turn ameliorates the sleep quality, life quality, and anti-oxidative functions in patients with sleep disorder.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 20-80 years old
2. Sleeping disorder patients with not or with low arousal threshold obstructive sleep apnea that were diagnosed by the doctor after PSG examination.

Exclusion Criteria:

1. Chronic diseases: liver, renal, gastrointestinal, cardiovascular diseases
2. Cancer
3. Pregnant
4. Be allergy to the intervention materials or having supplements /drugs which might affect the study outcome.

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2022-11-18 (Actual); Primary Completion 2023-12-18 (Actual); Study Completion 2023-12-18 (Actual)

PRIMARY OUTCOMES:
Change from Baseline The Pittsburgh Sleep Quality Index (PSQI) at two months | At the start of the experiment and at the 8th, 11th and 19th week
  PSQI is used to evaluate sleeping quality. A self-rated questionnaire which assesses sleep quality and disturbances over a 1-month time interval.
Change from Baseline Epworth Sleepiness Scale (ESS) at two months | At the start of the experiment and at the 8th, 11th and 19th week
  ESS i a self-administered questionnaire, and is used to assess the 'daytime sleepiness' of the patients.
Change from Baseline Beck Depression Inventory-II (BDI-11) score at two months | At the start of the experiment and at the 8th, 11th and 19th week
  BDI-11 is a self-report questionnaire rating measurements characteristic attitudes and symptoms of depression.
Change from Baseline Beck Anxiety Inventory (BAI) score at two months | At the start of the experiment and at the 8th, 11th and 19th week
  BAI is a self-report questionnaire that is used for measuring the severity of anxiety.
Change from Baseline Short form-12 items health survey (SF-12) at two months | At the start of the experiment and at the 8th, 11th and 19th week
  SF-12 is a general health questionnaire, which evaluated quality of life.

SECONDARY OUTCOMES:
Anthropometric assessmrnt | At the start of the experiment and at the 4th, 8th, 11th, 15th and 19th week
  BMI (kg/m^2), body composition and blood pressure (mmHg)
Liver function | At the start of the experiment and at the 8th, 11th and 19th week
  Serum AST and ALT (U/L)
Kidney function | At the start of the experiment and at the 8th, 11th and 19th week
  Serum BUN (mg/dL),Creatinine (mg/dL), eGFR (mL/min) and urine acid (mg/dL)
Lipid profile | At the start of the experiment and at the 8th, 11th and 19th week
  Serum HDL-C, LDL-C, triglyceride and total cholesterol (mg/dL)
Hematology | At the start of the experiment and at the 8th, 11th and 19th week
  WBC (10^3/uL), RBC (10^6/uL), hemoglobin (g/dL), hematocrit (%), MCV(fL), MCH (pg), MCHC (g/dL), platelet (10^3/uL), neutrophils (%), lymphocytes (%), monocytes (%), eosinophils (%) and basophils(%).
Antioxidative status | At the start of the experiment and at the 8th, 11th and 19th week
  Concentration of thiobarbituric acid-reactive substance, glutathione/oxidized glutathione ratio
Sesamin and it's metabolite | At the start of the experiment and at the 8th, 11th and 19th week
  Concentration of serum sesamin and it's metabolite

CONTACTS AND LOCATIONS:
Locations (2):
- Taiwan (2):
  - Taipei Medical University-Shuang Ho Hospital,Ministry of Health and Welfare, New Taipei City
  - Taipei Medical University, Taipei